CLINICAL TRIAL: NCT03951987
Title: Investigation of the Pharmacokinetic Properties of CG5503 After 2 Minutes Intravenous Infusion With and Without Oral Coadministration of Charcoal in a Randomised, Open, Single Dose, 2-way Crossover, Phase I Study in 12 Healthy Male Volunteers
Brief Title: Investigation How CG5503 is Taken up and Excreted From the Body After 2 Minutes Intravenous Infusion With and Without Oral Co-administration of Charcoal
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HP5503/11
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Pharmacokinetic
MeSH Terms: interventions — Tapentadol

STUDY DESIGN:
Intervention Model Description: The randomization was in the ratio 1:1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A: 4 ml CG5503 (Experimental): 4 ml of the CG5503 i.v. infusion solution corresponding to 40 mg CG5503 (tapentadol hydrochloride) was administered as a 2 minutes infusion.
  Interventions: Drug: 4 ml CG5503
- Treatment B: 4 ml CG5503; 5 g charcoal powder (Experimental): 4 ml of the CG5503 i.v. infusion solution corresponding to 40 mg CG5503 (tapentadol hydrochloride) with oral co-administration of charcoal (5 g charcoal were co-administered orally at 1, 0.5 hours and 10 minutes before the start of CG5503 infusion and 0.5, 1, 1.5, 2 and 4 hours thereafter)
  Interventions: Drug: 4 ml CG5503; Drug: 5 g charcoal powder

INTERVENTIONS:
Drug: 4 ml CG5503 — 4 ml of the CG5503 infusion solution corresponding to 40 mg CG5503 (tapentadol hydrochloride).
Drug: 5 g charcoal powder — Oral administration of 5 g charcoal powder suspended in 100 ml tap water.
  Other Names: Tradename: Kohle-Pulvis Pulver
  Arms: Treatment B: 4 ml CG5503; 5 g charcoal powder

SUMMARY:
This was a Phase I study in 12 healthy male participants to compare the pharmacokinetic properties of CG5503 (how it is taken up and excreted from the body) after 2 minutes intravenous (i.v.) infusion with and without oral co-administration of charcoal to investigate a potential gastrointestinal secretion of CG5503.

During the course of the study each participant received two infusions of 40 mg CG5503 without (treatment A) and with (treatment B) oral co-administration of charcoal. In treatment B, eight doses of 5 grams charcoal powder were co-administered orally at defined time points. The wash out phases were to be at least 4 to 14 days between the treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Male Caucasian participants aged 18 - 65 years.
* Body mass index (BMI) between 20 and 30 kilograms/square meter inclusive.
* Participants must be in good health as determined by medical history, physical examination, 12-lead electrocardiogram, vital signs, and clinical laboratory parameters (serum/urine biochemistry, serology and haematology). Minor deviations of laboratory values from the normal range may be accepted, if judged by the investigator to have no clinical relevance and if not considered to interfere with the study objectives.
* Negative human immunodeficiency virus (HIV)-1/-2 antibodies, hepatitis B surface (HBs)-antigen, hepatitis B core (HBc)-antibodies, hepatitis C virus (HCV)-antibodies at the screening examination.
* Participants giving written consent to participate within this trial.

Exclusion Criteria:

* Use of any medication within four weeks prior to commencement of the study (self-medication or prescription), if not on a stable basis.
* Diseases and functional disorders of the gastrointestinal tract, liver, cardiovascular system or kidneys.
* Malignancy.
* History of orthostatic hypotension.
* Resting pulse rate equal to or below 45 beats/min or equal to or above 100 beats/min.
* Systolic blood pressure equal to or below 100 mmHg or equal to or above 160 mmHg.
* Diastolic blood pressure equal to or below 50 mmHg or equal to or above 95 mmHg.
* Clinically relevant deviations in laboratory parameters.
* Drug allergy.
* Bronchial asthma.
* Participation in another clinical study in the last three months before starting this study (exception: characterization of metabolizer status).
* Blood donation (more than 100 milliliter) in the last three months before the start of the study.
* Evidence of alcohol or drug abuse.
* Positive drug abuse screening test.
* Extremely unbalanced diet (in the opinion of the investigator).
* Excessive consumption of food or beverages containing caffeine (more than five cups of coffee per day or other equivalent amounts of caffeine).
* Consumption of grapefruit juice two weeks before the start of the study.
* Known or suspected of not being able to comply with the study protocol.
* Not able to communicate meaningfully with the investigator and staff.
* Neurotic personality, psychiatric illness, or suicide risk.
* History of seizures or at risk (i.e. head trauma, epilepsy in family anamnesis, unclear loss of consciousness).

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2004-02 (Actual); Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter Serum: area under the concentration-time curve extrapolated to infinity (AUC0-inf) for CG5503 base | Pre-dose and up to 23 hours post-dose
  26 PK blood samples were obtained from each participant. Serum concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The AUC0-inf was calculated based on serum concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Saliva: area under the concentration-time curve extrapolated to infinity (AUC0-inf) for CG5503 base | Pre-dose and up to 23 hours post-dose
  16 PK saliva samples were obtained from each participant. Saliva concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. Participants were asked to donate saliva as much as possible in approximately 0.5 minutes. The AUC0-inf was calculated based on saliva concentration-time data (using the actual saliva sampling time intervals).
Pharmacokinetic parameter Serum: area under the concentration-time curve extrapolated to infinity (AUC0-inf) for CG5503-glucuronide | Pre-dose and up to 23 hours post-dose
  26 PK blood samples were obtained from each participant. Serum concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The AUC0-inf was calculated based on serum concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Serum: area under the concentration-time curve extrapolated to infinity (AUC0-inf) for CG5503-sulphate | Pre-dose and up to 23 hours post-dose
  26 PK blood samples were obtained from each participant. Serum concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The AUC0-inf was calculated based on serum concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Serum: area under the concentration-time curve from 0 to time t (AUC0-t) for CG5503 base | Pre-dose and up to 23 hours post-dose
  26 PK blood samples were obtained from each participant. Serum concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The AUC0-t was calculated based on serum concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Saliva: area under the concentration-time curve from 0 to time t (AUC0-t) for CG5503 base | Pre-dose and up to 23 hours post-dose
  16 PK saliva samples were obtained from each participant. Saliva concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. Participants were asked to donate saliva as much as possible in approximately 0.5 minutes. The AUC0-t was calculated based on saliva concentration-time data (using the actual saliva sampling time intervals).
Pharmacokinetic parameter Serum: area under the concentration-time curve from 0 to time t (AUC0-t) for CG5503-glucuronide | Pre-dose and up to 23 hours post-dose
  26 PK blood samples were obtained from each participant. Serum concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The AUC0-t was calculated based on serum concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Serum: area under the concentration-time curve from 0 to time t (AUC0-t) for CG5503-sulphate | Pre-dose and up to 23 hours post-dose
  26 PK blood samples were obtained from each participant. Serum concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The AUC0-t was calculated based on serum concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Serum: maximum concentration (Cmax) for CG5503 base | Pre-dose and up to 23 hours post-dose
  26 PK blood samples were obtained from each participant. Serum concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The Cmax was calculated based on serum concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Saliva: maximum concentration (Cmax) for CG5503 base | Pre-dose and up to 23 hours post-dose
  16 PK saliva samples were obtained from each participant. Saliva concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. Participants were asked to donate saliva as much as possible in approximately 0.5 minutes. tubes. The Cmax was calculated based on saliva concentration-time data (using the actual saliva sampling time intervals).
Pharmacokinetic parameter Serum: maximum concentration (Cmax) for CG5503-glucuronide | Pre-dose and up to 23 hours post-dose
  26 PK blood samples were obtained from each participant. Serum concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The Cmax was calculated based on serum concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Serum: maximum concentration (Cmax) for CG5503-sulphate | Pre-dose and up to 23 hours post-dose
  26 PK blood samples were obtained from each participant. Serum concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The Cmax was calculated based on serum concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Serum: time to maximum concentration (tmax) for CG5503 base | Pre-dose and up to 23 hours post-dose
  26 PK blood samples were obtained from each participant. Serum concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The tmax was calculated based on serum concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Saliva: time to maximum concentration (tmax) for CG5503 base | Pre-dose and up to 23 hours post-dose
  16 PK saliva samples were obtained from each participant. Saliva concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. Participants were asked to donate saliva as much as possible in approximately 0.5 minutes. The tmax was calculated based on saliva concentration-time data (using the actual saliva sampling time intervals).
Pharmacokinetic parameter Serum: time to maximum concentration (tmax) for CG5503-glucuronide | Pre-dose and up to 23 hours post-dose
  26 PK blood samples were obtained from each participant. Serum concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The tmax was calculated based on serum concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Serum: time to maximum concentration (tmax) for CG5503-sulphate | Pre-dose and up to 23 hours post-dose
  26 PK blood samples were obtained from each participant. Serum concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The tmax was calculated based on serum concentration-time data (using the actual blood sampling times).

SECONDARY OUTCOMES:
Pharmacokinetic parameter Serum: extrapolated AUC expressed as a percentage of total AUC0-inf (AUC%extr) for CG5503 base | Pre-dose and up to 23 hours post-dose
  26 PK blood samples were obtained from each participant. Serum concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The AUC%extr was calculated based on serum concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Saliva: extrapolated AUC expressed as a percentage of total AUC0-inf (AUC%extr) for CG5503 base | Pre-dose and up to 23 hours post-dose
  16 PK saliva samples were obtained from each participant. Saliva concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. Participants were asked to donate saliva as much as possible in approximately 0.5 minutes. The AUC%extr was calculated based on saliva concentration-time data (using the actual saliva sampling time intervals).
Pharmacokinetic parameter Serum: extrapolated AUC expressed as a percentage of total AUC0-inf (AUC%extr) for CG5503-glucuronide | Pre-dose and up to 23 hours post-dose
  26 PK blood samples were obtained from each participant. Serum concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The AUC%extr was calculated based on serum concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Serum: extrapolated AUC expressed as a percentage of total AUC0-inf (AUC%extr) for CG5503-sulphate | Pre-dose and up to 23 hours post-dose
  26 PK blood samples were obtained from each participant. Serum concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The AUC%extr was calculated based on serum concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Serum: apparent terminal elimination rate constant (λz) for CG5503 base | Pre-dose and up to 23 hours post-dose
  26 PK blood samples were obtained from each participant. Serum concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The λz was calculated based on serum concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Saliva: apparent terminal elimination rate constant (λz) for CG5503 base | Pre-dose and up to 23 hours post-dose
  16 PK saliva samples were obtained from each participant. Saliva concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. Participants were asked to donate saliva as much as possible in approximately 0.5 minutes. The λz was calculated based on saliva concentration-time data (using the actual saliva sampling time intervals).
Pharmacokinetic parameter Serum: apparent terminal elimination rate constant (λz) for CG5503-glucuronide | Pre-dose and up to 23 hours post-dose
  26 PK blood samples were obtained from each participant. Serum concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The λz was calculated based on serum concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Serum: apparent terminal elimination rate constant (λz) for CG5503-sulphate | Pre-dose and up to 23 hours post-dose
  26 PK blood samples were obtained from each participant. Serum concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The λz was calculated based on serum concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Serum: the apparent half-life associated with the terminal elimination phase (t1/2,z) for CG5503 base | Pre-dose and up to 23 hours post-dose
  26 PK blood samples were obtained from each participant. Serum concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The t½z was calculated based on serum concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Saliva: the apparent half-life associated with the terminal elimination phase (t1/2,z) for CG5503 base | Pre-dose and up to 23 hours post-dose
  16 PK saliva samples were obtained from each participant. Saliva concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. Participants were asked to donate saliva as much as possible in approximately 0.5 minutes. The t½z was calculated based on saliva concentration-time data (using the actual saliva sampling time intervals).
Pharmacokinetic parameter Serum: the apparent half-life associated with the terminal elimination phase (t1/2,z) for CG5503-glucuronide | Pre-dose and up to 23 hours post-dose
  26 PK blood samples were obtained from each participant. Serum concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The t½z was calculated based on serum concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Serum: the apparent half-life associated with the terminal elimination phase (t1/2,z) for CG5503-sulphate | Pre-dose and up to 23 hours post-dose
  26 PK blood samples were obtained from each participant. Serum concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The t½z was calculated based on serum concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Serum: total serum or blood clearance of drug after intravenous administration (CL) for CG5503 base | Pre-dose and up to 23 hours post-dose
  26 PK blood samples were obtained from each participant. Serum concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The CL was calculated based on serum concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Saliva: total clearance of drug after intravenous administration (CL) for CG5503 base | Pre-dose and up to 23 hours post-dose
  16 PK saliva samples were obtained from each participant. Saliva concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. Participants were asked to donate saliva as much as possible in approximately 0.5 minutes. The CL was calculated based on saliva concentration-time data (using the actual saliva sampling time intervals).
Pharmacokinetic parameter Serum: total serum or blood clearance of drug after intravenous administration (CL) for CG5503-glucuronide | Pre-dose and up to 23 hours post-dose
  26 PK blood samples were obtained from each participant. Serum concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The CL was calculated based on serum concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Serum: total serum or blood clearance of drug after intravenous administration (CL) for CG5503-sulphate | Pre-dose and up to 23 hours post-dose
  26 PK blood samples were obtained from each participant. Serum concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The CL was calculated based on serum concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Serum: the apparent volume of distribution associated with terminal phase after intravenous administration (Vz) for CG5503 base | Pre-dose and up to 23 hours post-dose
  26 PK blood samples were obtained from each participant. Serum concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The Vz was calculated based on serum concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Saliva: the apparent volume of distribution associated with terminal phase after intravenous administration (Vz) for CG5503 base | Pre-dose and up to 23 hours post-dose
  16 PK saliva samples were obtained from each participant. Saliva concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. Participants were asked to donate saliva as much as possible in approximately 0.5 minutes. The Vz was calculated based on saliva concentration-time data (using the actual saliva sampling time intervals).
Pharmacokinetic parameter Serum: the apparent volume of distribution associated with terminal phase after intravenous administration (Vz) for CG5503-glucuronide | Pre-dose and up to 23 hours post-dose
  26 PK blood samples were obtained from each participant. Serum concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The Vz was calculated based on serum concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Serum: the apparent volume of distribution associated with terminal phase after intravenous administration (Vz) for CG5503-sulphate | Pre-dose and up to 23 hours post-dose
  26 PK blood samples were obtained from each participant. Serum concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The Vz was calculated based on serum concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Urine: renal excretion (Ae % of dose) for CG5503 base | Pre-dose and up to 23 hours post-dose
  12 PK urine samples were obtained from each participant. Urine concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The Ae (% of dose) was calculated based on urine concentration-time data (using the actual urine sampling time intervals).
Pharmacokinetic parameter Urine: renal excretion (Ae % of dose) for CG5503-glucuronide | Pre-dose and up to 23 hours post-dose
  12 PK urine samples were obtained from each participant. Urine concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The Ae (% of dose) was calculated based on urine concentration-time data (using the actual urine sampling time intervals).
Pharmacokinetic parameter Urine: renal excretion (Ae % of dose) for CG5503-sulphate | Pre-dose and up to 23 hours post-dose
  12 PK urine samples were obtained from each participant. Urine concentrations were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The Ae (% of dose) was calculated based on urine concentration-time data (using the actual urine sampling time intervals).

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (1):
- Department of Clinical Pharmacology Grünenthal GmbH, Aachen, Germany

IPD SHARING:
Plan to Share IPD: No